CLINICAL TRIAL: NCT02271425
Title: An Absolute Bioavailability Study of Evacetrapib in Healthy Subjects Using the Intravenous Tracer Method
Brief Title: A Study to Measure the Amount of Evacetrapib That Enters the Blood Stream in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14622; I1V-MC-EIAT (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evacetrapib Tablet + Evacetrapib Intravenous (Experimental): A single oral dose of 130 milligrams (mg) evacetrapib tablet + a single intravenous (IV) dose of 175 micrograms (μg)[¹³C₈] evacetrapib administered over a 4 hour infusion.
  Interventions: Drug: Evacetrapib Tablet; Drug: Evacetrapib Intravenous

INTERVENTIONS:
Drug: Evacetrapib Tablet — Oral administration
  Other Names: LY2484595
Drug: Evacetrapib Intravenous — Intravenous administration
  Other Names: LY2484595

SUMMARY:
Evacetrapib (study drug) is an investigational drug being developed with the aim to help people at high risk of heart problems in the future.

In this study we will be comparing how much of the study drug gets into the blood stream when it is given as a single dose (in tablet form) compared to an intravenous injection (given directly into a vein via a small needle).

The study is expected to last at least 15 days for each participant, not including screening. Screening will occur up to 28 days before the study drug is given.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination
* Female participants are post menopausal women or women not of child bearing potential due to surgical sterilization (at least 6 weeks after surgical hysterectomy, bilateral oophorectomy, or tubal occlusion) confirmed by medical history, or menopause
* Have a body mass index (BMI) of less than 32 kilograms per square meter (kg/m^2)
* Have given written informed consent approved by Eli Lilly and Company and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Have known allergies to evacetrapib, related compounds or any components of the formulation, intolerance to alcohol containing products, or history of significant allergic disease as determined by the investigator
* Have an abnormal blood pressure as determined by the investigator
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Are women who are pregnant or are lactating
* Have used or intend to use over-the-counter or prescription medications (including vitamins/mineral supplements/herbal medicine) 14 days prior to the first dose and during the study. The use of topical medicine, provided there is no evidence of chronic dosing with risk of systemic exposure, and occasional acetaminophen is acceptable
* Have donated blood of more than 500 milliliter (mL) within the last 3 months
* Are unwilling to comply with the dietary requirements/restrictions during the study:

  * Consume only the meals provided during the inpatient appointments,
  * Refrain from eating any food or drinking any beverages containing grapefruit, grapefruit juice, Seville oranges, Seville orange juice, star fruit, pomelo, or commercial apple juice or orange juice for at least 7 days prior to the first dose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Evacetrapib Tablet + Evacetrapib Intravenous: Single oral dose of 130 milligrams (mg) evacetrapib tablet + a single intravenous (IV) dose of 175 micrograms (μg)[¹³C₈] evacetrapib administered over a 4 hour infusion.
Period: Overall Study
Arm/Group | Evacetrapib Tablet + Evacetrapib Intravenous
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Evacetrapib Tablet + Evacetrapib Intravenous: Single oral dose of 130 mg evacetrapib tablet + a single IV dose of 175 µg [¹³C₈] evacetrapib administered over a 4 hour infusion.
Arm/Group | Evacetrapib Tablet + Evacetrapib Intravenous
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Dose Normalized Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Evacetrapib
Time Frame: Day 1:Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.25, 4.5, 5, 5.5, 6, 6.5, 8, 10, 12, Day 2; 24, 36 Day 3; 48 Day 4; 72 Day 5; 96 Day 6; 120 Day 7; 144 and Day 8; 168 hours post-dose
Population: All participants who received at least one dose of study drug and had evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogramxhour/milliliter/mg (ngxh/ml/mg)
Groups:
- Evacetrapib: Tablet: A single oral dose of 130 mg evacetrapib tablet
- Evacetrapib: Intravenous: A single IV dose of 175 μg [¹³C₈] evacetrapib administered over a 4 hour infusion.
Arm/Group | Evacetrapib: Tablet | Evacetrapib: Intravenous
Number analyzed (Participants) | 8 | 8
nanogramxhour/milliliter/mg (ngxh/ml/mg) | 111 (21) | 248 (16)

ADVERSE EVENTS:
Description: The adverse events were collected from participants who received simultaneous administration of a single oral dose and a 4-hour intravenous (IV) infusion.
Arm/Group | Evacetrapib Tablet + Evacetrapib Intravenous
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib Tablet + Evacetrapib Intravenous (N=8)
Catheter site pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days